CLINICAL TRIAL: NCT07220902
Title: Levetiracetam Compared to Magnesium Sulfate for Prevention of Eclamptic Seizure: A Randomized Controlled Trial "LEVMag Trial"
Brief Title: Levetiracetam Compared to Magnesium Sulfate for Prevention of Eclamptic Seizure
Acronym: LEVMag
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nebraska Methodist Health System (Other)
Responsible Party: Principal Investigator, Todd Lovgren, Primary Investigator, Nebraska Methodist Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1559
Record Dates: First submitted 2025-10-20; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Severe Preeclampsia; Eclampsia Preeclampsia
Keywords: Seizure; Prophylaxis; Preeclampsia; Eclampsia; Keppra; Levetiracetam; Magnesium; LEVMag; Equivalence
MeSH Terms: conditions — Pre-Eclampsia; Seizures; Eclampsia | interventions — Levetiracetam; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levetiracetam Arm (Experimental): This experimental arm will receive oral levetiracetam 3 times daily after an initial loading oral dose.
  Interventions: Drug: Levetiracetam
- Magnesium Sulfate Arm (Active Comparator): This arm will receive standard treatment- a loading dose of magnesium sulfate followed by a continuous infusion that is the current standard of care (4 gram bolus followed by 2grams per hour continuous infusion).
  Interventions: Drug: magnesium sulfate

INTERVENTIONS:
Drug: Levetiracetam — 1g oral loading dose followed by 300mg q 8 hours beginning 8 hours after loading dose.
  Other Names: Keppra
  Arms: Levetiracetam Arm
Drug: magnesium sulfate — 4gram bolus followed by 2g per hour continuous infusion
  Arms: Magnesium Sulfate Arm

SUMMARY:
The goal of this study is to compare levetiracetam to magnesium sulfate for the prevention of eclamptic seizures in pregnant persons with severe preeclampsia that are 32 or more weeks pregnant. This is an equivalence study so our primary goal is to see no difference in the incidence of seizure in the two groups. Since side effects can be a significant problem with magnesium sulfate and these patients are at significant risk of life threatening complications, we also plan to evaluate several secondary outcomes in the mothers and the babies, including:

severe allergic reaction, magnesium toxicity, ICU admission, hospital readmission, transfusion for any reason, pulmonary edema, cardiomyopathy, Posterior Reversible Encephalopathy Syndrome, eclamptic seizure, loss of vision, stroke, renal injury requiring dialysis, cardiac arrest, maternal death, unexpected stillbirth or neonatal death, NICU admission, Apgars and length of neonatal respiratory support.

DETAILED DESCRIPTION:
Levetiracetam Compared to Magnesium Sulfate for Prevention of Eclamptic Seizure: A Randomized Controlled Trial Study Protocol

1. Study Title: Levetiracetam Compared to Magnesium Sulfate for Prevention of Eclamptic Seizure: A Randomized Controlled Trial (LEVMag Trial)
2. Objectives

   * Primary Objective: To assess whether Levetiracetam is non-inferior to Magnesium Sulfate in preventing eclamptic seizures in laboring and postpartum women with severe preeclampsia and HELLP syndrome.
   * Secondary Objectives: To compare the safety profiles, maternal and neonatal outcomes, and incidence of adverse events between the two study medications.
3. Study Design

   * Design: Prospective, randomized, controlled, open-label, non-inferiority trial.
   * Setting: Single Urban Level III Obstetric Facility
   * Duration: 72-84 months (including recruitment, treatment, and follow-up).
4. Study Population

   * Inclusion Criteria:

     * Pregnant or postpartum women aged 19 years or older
     * Diagnosed with preeclampsia with severe features, superimposed preeclampsia or HELLP syndrome
     * At risk for eclampsia and eligible for seizure prophylaxis
     * Less than 2 hours exposure to magnesium sulfate or greater than 48 hours since last dose.
   * Exclusion Criteria:

     * <32 weeks estimated gestational age
     * History of epilepsy or seizure disorders unrelated to pregnancy
     * Allergy or contraindication to Levetiracetam or Magnesium Sulfate
     * Severe renal impairment (Oliguria <120ml in 4 hours)
     * Plan for neonatal comfort care
5. Intervention/Comparator

   * Intervention Arm: Levetiracetam 1g PO followed by Levetiracetam 1500 mg/day immediate release PO in 3 divided doses. Divided doses to begin 8 hours after initial 1g loading dose.
   * Control Arm: Magnesium Sulfate 4gm IV over 15-20min followed by 2gm/hr IV infusion (current hospital protocol).
6. Outcome Measures

   * Primary Outcome:

     o Incidence of eclamptic seizures from enrollment to discharge from delivery hospitalization.
   * Secondary Outcomes:

     * Composite outcome of adverse events and severe adverse events
     * Neonatal 1 and 5 minute Apgar scores, NICU admission, length of respiratory support, neonatal death and stillbirth
7. Sample Size and Power Calculation

   • Assumptions:
   * Expected seizure incidence with Magnesium Sulfate: 0.5%
   * Non-inferiority margin: 1%
   * Power: 80%
   * Alpha: 0.05 (one-sided)
   * Sample size per group: 620
   * Total sample size: 1,240
8. Randomization Technique

   • Permuted randomization scheme will be used.
   * Participants will be randomized 1:1 using a computer-generated randomization tool.
   * Block randomization with variable block sizes (4,6,8) will ensure balance between groups.
   * Allocation concealment will be maintained using sealed, opaque envelopes.
9. Enrollment

   * We are collaborating with the Pharmacy Department to improve timing of patient enrollment. In addition to trained research nurses, participating Pharmacists will be CITI certified.
   * Patients will be identified when an order is entered for Magnesium Sulfate for seizure prophylaxis. A research pharmacist, research RN or principal investigator will then review the chart to ensure the patient meets study inclusion criteria.
   * For patients that meet inclusion criteria they will be approached in the location they are receiving care to review consent forms and be provided the patient bill of rights.
   * Those choosing to participate and completing the consent process will then be randomized. The next randomization envelope will be opened to determine their assigned treatment group and pharmacist will enter the appropriate orders.
   * Due to the urgent nature of this treatment, our goal is to complete enrollment and study assignment in sixty minutes or less after the initial order is received.
10. Adverse Event Reporting

    * Adverse events (AEs) and serious adverse events (SAEs) will be recorded and reported in accordance with ICH-GCP guidelines (see below).
    * SAEs will be reported to the IRB and Data Safety Monitoring Board (DSMB) within 24 hours of when they are identified.
    * Interim safety analyses will be performed by the DSMB every 300 enrolled patients.
    * DSMB- 1 outside MFM provider, 1 non PI Methodist MFM, 1 Methodist OB provider.
11. Ethical Considerations and Informed Consent

    * Approval will be obtained from the Institutional Review Board (IRB) and registered with clinicaltrials.gov once IRB approval is attained.
    * Participants will be provided with a detailed informed consent form outlining study procedures, risks, and rights.

Study Justification and Protocol Clarifications Modern anti-epileptic drugs have not been evaluated in their ability to prevent eclamptic seizures. The last studies comparing magnesium sulfate were performed against Nimodipine, a calcium channel blocker, over 20 years ago and phenytoin around 30 years ago. Magnesium sulfate is the current gold standard for seizure prophylaxis in women with hypertensive disease of pregnancy. It is a high risk medication that requires careful management and titration due to the risk for toxicity, respiratory depression, cardiac arrhythmia and death. Despite the high risk nature of a magnesium drip there has not been recent effort to identify safer medications for the prevention of eclamptic seizures. The study authors advocate for the study of Levetiracetam commercially known as Keppra®.

Levetiracetam is FDA approved for tonic-clonic seizures and is already used during pregnancy with an excellent safety profile in women with epilepsy (see appendix A). Use in this trial would be short term (likely 36-96 hours) and in late preterm or term pregnancies. This poses no risk for fetal malformation or birth defects as organogenesis is completed by 12 weeks and the study will enroll patients after 32 weeks gestation. As noted, levetiracetam has demonstrated safety in pregnancy in women with epilepsy and is safe in women who are breastfeeding. It has few significant complications specific to the medication itself and the short-term nature of the use in this study further mitigates those risks. Immediate release levetiracetam reaches maximum concentration in the blood in approximately 1 hour. Magnesium sulfate reaches a peak in 30 minutes when a bolus is given with levels falling by 60 minutes to roughly 2x physiologic levels, but typically below the 2mmol/L that is academically thought to be therapeutic. There is no currently established therapeutic dose based on scientific data. It is not recommended to routinely check magnesium levels during infusion unless there is concern for toxicity or renal impairment.

Inclusion/Exclusion - the reasoning behind our various criteria are related to state law, drug metabolism and to prevent confounders. Patients under 32 weeks gestation are excluded as they should receive magnesium sulfate for fetal neuroprotection and this exposure would confound the exposure groups, 19 y/o is the age of consent in Nebraska and renal impairment is important as both magnesium sulfate and levetiracetam are renally cleared. Since magnesium is rapidly cleared from the body we are choosing to include patients with less than 2 hours of exposure to magnesium or who have not received magnesium in the last 48 hours as we feel this does not clinically confound results due to short duration of exposure or complete clearance of the medication after prior exposure.

Dosing for magnesium is based on medically standardized protocol and Levetiracetam dosing is based on adult dosing in non-pregnant individuals with tonic-clonic seizures.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or postpartum women aged 19 years or older
* Diagnosed with preeclampsia with severe features, superimposed preeclampsia or HELLP syndrome
* At risk for eclampsia and eligible for seizure prophylaxis
* Less than 2 hours exposure to magnesium sulfate or greater than 48 hours since last dose.
* Admitted or plan to proceed with delivery

Exclusion Criteria:

* <32 weeks estimated gestational age
* History of epilepsy or seizure disorders unrelated to pregnancy
* Allergy or contraindication to Levetiracetam or Magnesium Sulfate
* Severe renal impairment (Oliguria <120ml in 4 hours)
* Plan for neonatal comfort care

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Birthing persons are the only population that can be included as the study is being conducted in pregnancy.
Enrollment: 1240 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2033-12-31 (Estimated); Study Completion 2034-07 (Estimated)

PRIMARY OUTCOMES:
Eclamptic Seizure | From enrollment until then end of monitoring at 6 weeks postpartum.
  Seizure based on clinical diagnosis by managing physician. It will be considered and eclamptic seizure for purposes of the study if it occurs following enrollment in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Lovgren, MD, Principal Investigator — Nebraska Methodist Health System
Locations (1):
- Methodist Women's Hospital, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared on a case-by-case basis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be shared beginning 1 year after publication.
Access Criteria: Deidentified IPD will be shared on a case by case basis with principal investigators by contacting the PI for this study.

REFERENCES:
- [Background] Johannessen Landmark C, Patsalos PN. Drug interactions involving the new second- and third-generation antiepileptic drugs. Expert Rev Neurother. 2010 Jan;10(1):119-40. doi: 10.1586/ern.09.136. PMID 20021326
- [Background] Loscher W, Schmidt D. New Horizons in the development of antiepileptic drugs: Innovative strategies. Epilepsy Res. 2006 Jun;69(3):183-272. doi: 10.1016/j.eplepsyres.2006.03.014. PMID 16835945
- [Background] Perucca P, Gilliam FG. Adverse effects of antiepileptic drugs. Lancet Neurol. 2012 Sep;11(9):792-802. doi: 10.1016/S1474-4422(12)70153-9. Epub 2012 Jul 24. PMID 22832500
- [Background] French JA, Kanner AM, Bautista J, Abou-Khalil B, Browne T, Harden CL, Theodore WH, Bazil C, Stern J, Schachter SC, Bergen D, Hirtz D, Montouris GD, Nespeca M, Gidal B, Marks WJ Jr, Turk WR, Fischer JH, Bourgeois B, Wilner A, Faught RE Jr, Sachdeo RC, Beydoun A, Glauser TA; American Academy of Neurology Therapeutics and Technology Assessment Subcommittee; American Academy of Neurology Quality Standards Subcommittee; American Epilepsy Society Quality Standards Subcommittee; American Epilepsy Society Therapeutics and Technology Assessment Subcommittee. Efficacy and tolerability of the new antiepileptic drugs, I: Treatment of new-onset epilepsy: report of the TTA and QSS Subcommittees of the American Academy of Neurology and the American Epilepsy Society. Epilepsia. 2004 May;45(5):401-9. doi: 10.1111/j.0013-9580.2004.06204.x. PMID 15101821
- [Background] Patsalos PN. Clinical pharmacokinetics of levetiracetam. Clin Pharmacokinet. 2004;43(11):707-24. doi: 10.2165/00003088-200443110-00002. PMID 15301575
- [Background] Kanner AM, Ashman E, Gloss D, Harden C, Bourgeois B, Bautista JF, Abou-Khalil B, Burakgazi-Dalkilic E, Llanas Park E, Stern J, Hirtz D, Nespeca M, Gidal B, Faught E, French J. Practice guideline update summary: Efficacy and tolerability of the new antiepileptic drugs I: Treatment of new-onset epilepsy: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology and the American Epilepsy Society. Neurology. 2018 Jul 10;91(2):74-81. doi: 10.1212/WNL.0000000000005755. Epub 2018 Jun 13. PMID 29898971
- [Background] Appleton RE, Rainford NE, Gamble C, Messahel S, Humphreys A, Hickey H, Woolfall K, Roper L, Noblet J, Lee E, Potter S, Tate P, Al Najjar N, Iyer A, Evans V, Lyttle MD. Levetiracetam as an alternative to phenytoin for second-line emergency treatment of children with convulsive status epilepticus: the EcLiPSE RCT. Health Technol Assess. 2020 Nov;24(58):1-96. doi: 10.3310/hta24580. PMID 33190679
- [Background] Shorvon SD, Lowenthal A, Janz D, Bielen E, Loiseau P. Multicenter double-blind, randomized, placebo-controlled trial of levetiracetam as add-on therapy in patients with refractory partial seizures. European Levetiracetam Study Group. Epilepsia. 2000 Sep;41(9):1179-86. doi: 10.1111/j.1528-1157.2000.tb00323.x. PMID 10999557
- [Background] Ben-Menachem E, Falter U. Efficacy and tolerability of levetiracetam 3000 mg/d in patients with refractory partial seizures: a multicenter, double-blind, responder-selected study evaluating monotherapy. European Levetiracetam Study Group. Epilepsia. 2000 Oct;41(10):1276-83. doi: 10.1111/j.1528-1157.2000.tb04605.x. PMID 11051122
- [Background] Chamberlain JM, Kapur J, Shinnar S, Elm J, Holsti M, Babcock L, Rogers A, Barsan W, Cloyd J, Lowenstein D, Bleck TP, Conwit R, Meinzer C, Cock H, Fountain NB, Underwood E, Connor JT, Silbergleit R; Neurological Emergencies Treatment Trials; Pediatric Emergency Care Applied Research Network investigators. Efficacy of levetiracetam, fosphenytoin, and valproate for established status epilepticus by age group (ESETT): a double-blind, responsive-adaptive, randomised controlled trial. Lancet. 2020 Apr 11;395(10231):1217-1224. doi: 10.1016/S0140-6736(20)30611-5. Epub 2020 Mar 20. PMID 32203691
- [Background] Hope OA, Harris KM. Management of epilepsy during pregnancy and lactation. BMJ. 2023 Sep 8;382:e074630. doi: 10.1136/bmj-2022-074630. PMID 37684052
- [Background] Carosella CM, Johnson EL. Special Issues in Medical Management: Hormones and Pregnancy in Epilepsy. Semin Neurol. 2025 Apr;45(2):198-205. doi: 10.1055/a-2551-0688. Epub 2025 Apr 3. PMID 40179957
- [Background] Tomson T, Battino D, Bonizzoni E, Craig J, Lindhout D, Perucca E, Sabers A, Thomas SV, Vajda F; EURAP Study Group. Comparative risk of major congenital malformations with eight different antiepileptic drugs: a prospective cohort study of the EURAP registry. Lancet Neurol. 2018 Jun;17(6):530-538. doi: 10.1016/S1474-4422(18)30107-8. Epub 2018 Apr 18. PMID 29680205
- [Background] Meador KJ, Pennell PB, Harden CL, Gordon JC, Tomson T, Kaplan PW, Holmes GL, French JA, Hauser WA, Wells PG, Cramer JA; HOPE Work Group. Pregnancy registries in epilepsy: a consensus statement on health outcomes. Neurology. 2008 Sep 30;71(14):1109-17. doi: 10.1212/01.wnl.0000316199.92256.af. Epub 2008 Aug 13. PMID 18703463
- [Background] Mawhinney E, Craig J, Morrow J, Russell A, Smithson WH, Parsons L, Morrison PJ, Liggan B, Irwin B, Delanty N, Hunt SJ. Levetiracetam in pregnancy: results from the UK and Ireland epilepsy and pregnancy registers. Neurology. 2013 Jan 22;80(4):400-5. doi: 10.1212/WNL.0b013e31827f0874. Epub 2013 Jan 9. PMID 23303847
- [Background] Shallcross R, Bromley RL, Cheyne CP, Garcia-Finana M, Irwin B, Morrow J, Baker GA; Liverpool and Manchester Neurodevelopment Group; UK Epilepsy and Pregnancy Register. In utero exposure to levetiracetam vs valproate: development and language at 3 years of age. Neurology. 2014 Jan 21;82(3):213-21. doi: 10.1212/WNL.0000000000000030. Epub 2014 Jan 8. PMID 24401687
- [Background] Shallcross R, Bromley RL, Irwin B, Bonnett LJ, Morrow J, Baker GA; Liverpool Manchester Neurodevelopment Group; UK Epilepsy and Pregnancy Register. Child development following in utero exposure: levetiracetam vs sodium valproate. Neurology. 2011 Jan 25;76(4):383-9. doi: 10.1212/WNL.0b013e3182088297. PMID 21263139
- [Background] Chaudhry SA, Jong G, Koren G. The fetal safety of Levetiracetam: a systematic review. Reprod Toxicol. 2014 Jul;46:40-5. doi: 10.1016/j.reprotox.2014.02.004. Epub 2014 Mar 3. PMID 24602560